CLINICAL TRIAL: NCT02925741
Title: Clinical Trial of Silk-Like Linens for Prevention of Unit-Acquired Pressure Ulcers
Brief Title: Silk-Like Bed Linens for Prevention of Unit-Acquired Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Standard Textile (Unknown); Precision Fabrics Group, Inc. (Other)
Responsible Party: Principal Investigator, Mary Montague, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-752
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Pressure Ulcer
Keywords: bed linens
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Of 5 Medical ICUs at 1 quaternary care medical center, patients were assigned to groups based on bed availability by personnel who were blinded to linens used on those units.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silk-Like Linens (Experimental): Patients in the experimental arm will be cared for on silk-like bed linens.
  Interventions: Other: Silk-Like Linens
- Standard Cotton Linens (No Intervention): Patients in the standard of care arm will be cared for on standard cotton bed linens.

INTERVENTIONS:
Other: Silk-Like Linens — Synthetic moisture-wicking fabric
  Other Names: Dermatherapy
  Arms: Silk-Like Linens

SUMMARY:
This study will use a traditional parallel randomization design with patients in five medical intensive care units at the Cleveland Clinic to evaluate the efficacy of silk-like bed sheets and underpads for prevention of Unit-Acquired Pressure Ulcers (UAPU). Adult hospitalized patients in beds with standard bed linens versus those with silk-like linens will be compared for 1) rate of development of UAPU, 2) time to develop the first UAPU, and the maximum severity of any UAPU that develop. Bed linens will be changed per unit protocol. Patient characteristics will be summarized using frequencies and percentages for categorical factors and means, standard deviations, percentiles and median and range for continuous measures. For the primary outcome of unit-acquired pressure ulcer rate, generalized linear mixed models, assuming a Poisson distribution for the outcome, and unit length of stay as an offset will be used. For the time to event analysis, frailty models will be used to assess whether time to first pressure ulcer differs between treatment types. Generalized linear mixed models will be used for other secondary endpoints, including maximum severity of observed pressure ulcers

DETAILED DESCRIPTION:
Although there has been a large amount of research published on contributing factors to pressure ulcers, there has been little research related to the role that bed linens play in affecting moisture, friction, and shear that may lead to development of unit-acquired pressure ulcers (UAPU) for patients in acute care settings. This study will use a traditional parallel randomized design with patients in five medical intensive care units at the Cleveland Clinic to evaluate the efficacy of silk-like bed sheets and underpads for prevention of Unit-Acquired Pressure Ulcers (UAPU). Patients were randomly assigned by personnel who were blinded to the intervention based on bed availability. Nurses will assess all patients on standard bed linens and silk-like linens for development of UAPU. Adult hospitalized patients in beds with standard bed linens versus those with silk-like linens will be compared for 1) rate of development of UAPU, 2) time to develop the first UAPU, and the maximum severity of any UAPU that develop. Upon entry into the study, all patients will be assessed for baseline skin integrity by the admitting nurse. Demographic data (MRN; unit name; type of linen on bed; admitting diagnosis; dates of admission/discharge; age; gender; race; weight; Braden score; date, location, and stages of UAPU development; lab values (albumin, total protein); and categories of the Charlson Comorbidity Index will be recorded on data collection form by research nurse. Bed linens will be changed per unit protocol. A sample size of 3456 patients is estimated. Patient characteristics will be summarized using frequencies and percentages for categorical factors and means, standard deviations, percentiles and median and range for continuous measures. Comparisons of these patient characteristics, including Braden score, Charlson comorbidity index, unit length of stay and hospital length of stay, will be compared between linen types using generalized linear mixed effect models. For the primary outcome of unit-acquired pressure ulcer rate, generalized linear mixed models, assuming a Poisson distribution for the outcome, and unit length of stay as an offset will be used. In these models, linen type and study period will be used as fixed effects and each unit will be included as a random effect. For the time to event analysis, frailty models will be used to assess whether time to first pressure ulcer differs between treatment types. Generalized linear mixed models will be used for other secondary endpoints, including maximum severity of observed pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted into the medical intensive care unit during the one year study period

Exclusion Criteria:

* Patients who are transferred from one study unit to another study unit, data for their days on the second unit will be measured only if the second unit is in the same study arm as the sending unit
* Patients who are in the prone position
* Patients remaining on a unit past the two week washout period, will not be included in the crossover arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3343 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Montague, MSN, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven patients refused the synthetic linens.
Groups:
- Silk-like Linen: Patients being cared for on silk-like linens
- Standard Cotton Linen: Patients being cared for on standard cotton linens
Period: Overall Study
Arm/Group | Silk-like Linen | Standard Cotton Linen
Started | 1637 | 1706
Completed | 1626 | 1706
Not Completed | 11 | 0
Not completed — Withdrawal by Subject | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Silk-like Linen: Patients cared for on silk-like linen.
- Standard Cotton Linen: Patients cared for on standard cotton linen
- Total: Total of all reporting groups
Arm/Group | Silk-like Linen | Standard Cotton Linen | Total
Number analyzed (Participants) | 1626 | 1706 | 3332
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (16.6) | 60.3 (16.0) | 60.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not available for all subjects. Sex missing from 1 patient in the silk group and 1 patient in the cotton group.
  Participants
    number analyzed (Participants) | 1625 | 1705 | 3330
    Female | 769 | 796 | 1565
    Male | 856 | 909 | 1765
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 538 | 499 | 1037
  White | 1010 | 1104 | 2114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 78 | 103 | 181
Diagnostic Category [Count of Participants; unit: Participants] — Data not available for all subjects. Population: Data missing
  Participants
    number analyzed (Participants) | 1565 | 1611 | 3176
    Cardiovascular | 505 | 510 | 1015
    Gastrointestinal | 217 | 250 | 467
    Respiratory | 508 | 491 | 999
    Hematologic | 145 | 104 | 249
    Other | 190 | 256 | 446
Weight; kgs [Mean (Standard Deviation); unit: kgs] — Data not available for all subjects. Population: Data missing
  kgs
    number analyzed (Participants) | 1431 | 1480 | 2911
    (all) | 85.5 (29.7) | 85.4 (30.6) | 85.4 (30.1)
Albumin, mg/dL [Mean (Standard Deviation); unit: mg/dL] — Data not available for all subjects. Population: Data missing
  mg/dL
    number analyzed (Participants) | 1599 | 1706 | 3305
    (all) | 3.1 (0.71) | 3.0 (0.70) | 3.1 (0.70)
Total Protein, mg/dL [Mean (Standard Deviation); unit: mg/dL] — Data not available for all subjects. Population: Data missing
  mg/dL
    number analyzed (Participants) | 1599 | 1644 | 3243
    (all) | 6.2 (1.05) | 6.2 (1.01) | 6.2 (1.03)
Braden Score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Braden Scale is a valid and reliable tool which determines a patient's risk for developing a pressure ulcer. It consists of six individual subsets: sensory perception, moisture, activity, mobility, nutrition, and friction/shear. All subsets, with the exception of friction/shear are measured on a 1-4 scale; friction/shear measured on a 1-3 scale. The total score can range from 6 indicating a high risk of pressure injury development to 23 indicating low risk of pressure injury development. The level of risk dictates the intervention strategies that should be used.
  units on a scale | 15.5 (3.1) | 15.4 (3.1) | 15.4 (3.1)
APACHE [Mean (Standard Deviation); unit: calculated score (high= high acuity)] — APACHE II ("Acute Physiology And Chronic Health Evaluation II") is a severity-of-disease classification system, one of several ICU scoring systems. It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death Data not available for all subjects. Population: Missing data
  calculated score (high= high acuity)
    number analyzed (Participants) | 934 | 1064 | 1998
    (all) | 67.5 (28.7) | 66.4 (27.8) | 66.9 (28.2)
Admission Type [Count of Participants; unit: Participants] — Patient's location prior to MICU admission. Data not available for all subjects Population: Data missing
  Participants
    number analyzed (Participants) | 1623 | 1702 | 3325
    Outside | 460 | 484 | 944
    Emergency Department | 720 | 729 | 1449
    Direct Admission | 43 | 37 | 80
    Inpatient | 400 | 452 | 852
Charlson Comorbidity Index [Count of Participants; unit: Participants] — The categories are based on the sum of the weights. The categories are risk stratification groupings created by the instrument developer. There is a stepwise increase in the observed mortality with a higher comorbidity index, within each of the severity groups. Population: Data missing
  Participants
    number analyzed (Participants) | 1623 | 1704 | 3327
    0 | 309 | 282 | 591
    1-2 | 599 | 690 | 1289
    3-4 | 451 | 439 | 890
    5 or more | 264 | 293 | 557

OUTCOME MEASURES:

1. Primary Outcome: Rate of Development of Unit-acquired Pressure Ulcers
Description: Total count of the number of patients who developed unit acquired pressure ulcers during the study (count)
Time Frame: During MICU admission
Population: Total count and percentage of patients who developed a hospital acquired pressure injury (HAPI)
Measure: Count of Participants; unit: Participants
Groups:
- Silk-Like Linen: Patients in the experimental arm will be cared for on silk-like bed linens.
- Standard Cotton Linen: Patients in the control arm will be cared for on standard cotton linen.
Arm/Group | Silk-Like Linen | Standard Cotton Linen
Number analyzed (Participants) | 1626 | 1706
Participants | 45 | 42

2. Secondary Outcome: The Time to Develop the First Unit-acquired Pressure Ulcer
Description: The number of days spent in the intensive care unit prior to the development of a pressure ulcer
Time Frame: Days from admission to HAPI
Population: Number of days from admission to first HAPI for patients who developed a HAPI
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Silk-Like Linen: Patients in the experimental group will be cared for on silk-like linen.
- Standard Cotton Linen: Patients in the control group will be cared for on standard cotton linen.
Arm/Group | Silk-Like Linen | Standard Cotton Linen
Number analyzed (Participants) | 1626 | 1706
days | 6 [3 to 11] | 6 [3 to 10]

3. Secondary Outcome: Maximum Severity of Unit Acquired Pressure Injury (UAPI)
Description: HAPI staged by trained clinical nurses using the National Pressure Advisory Panel (NPUAP) staging definitions in which Stage 1 is the least severe with severity progressing through Stage 2, 3, 4, and unstageable. Unstageable is an evolving type of pressure injury evolving into a Stage 3 or 4.
Time Frame: During MICU admission
Population: For all patients, maximum stage of HAPI during medical intensive care unit (MICU) stay
Measure: Count of Participants; unit: Participants
Groups:
- Standard Cotton Linen: Patients in the control group were cared for on standard cotton linen.
Arm/Group | Silk-Like Linen | Standard Cotton Linen
Number analyzed (Participants) | 1626 | 1706
Participants
  Stage 1 | 6 | 9
  Stage 2-4 | 20 | 22
  Unstageable | 15 | 15
  No HAPI | 1585 | 1660

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Silk-like Linens; Standard Cotton Linens: This study will use a traditional parallel randomization design with patients in five medical intensive care units.
  Patients were assigned to groups based on bed availability by personnel who were blinded to linens used on those units. Each unit used the linens assigned by the randomization procedure for six months followed by a fourteen day washout period. Patient participation was based on the unit to which they were assigned.
Arm/Group | Silk-like Linens | Standard Cotton Linens
Serious Adverse Events (participants affected / at risk) | 0/1626 | 0/1706
Other Adverse Events (participants affected / at risk) | 2/1626 | 0/1706
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silk-like Linens (N=1626) | Standard Cotton Linens (N=1706)
CAUTI (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No